CLINICAL TRIAL: NCT04396821
Title: A Phase I/IIa Clinical Trial to Evaluate the Safety, Tolerability and Pharmacokinetics of TST001 Administered as Monotherapy or in Combination With Nivolumab or Standard of Care in Patients With Locally Advanced or Metastatic Solid Tumors
Brief Title: A Trial to Evaluate Safety and Tolerability of TST001 in Advanced or Metastatic Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Suzhou Transcenta Therapeutics Co., Ltd. (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TST001-1001
Record Dates: First submitted 2020-05-07; First posted 2020-05-21 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-11

CONDITIONS: Advanced Cancer; Gastric Cancer; Gastroesophageal-junction Cancer; Pancreatic Cancer
MeSH Terms: conditions — Stomach Neoplasms; Pancreatic Neoplasms | interventions — Nivolumab; Gemcitabine; Albumin-Bound Paclitaxel

STUDY DESIGN:
Intervention Model Description: Part A - 2 arms, Q2w and Q3w, 3+3 design dose escalation; Part B - dose expansion, 3 Cohorts
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Part A Q2W (Experimental): Dosed every 2 weeks IV with TST001, starting dose is 1 mg/kg, multiple dose levels will be tested.
  Interventions: Drug: TST001
- Part A Q3W (Experimental): Dosed every 3 weeks IV with TST001, starting dose is 3 mg/kg, and multiple dose levels will be tested.
  Interventions: Drug: TST001
- Part B Cohort A (Experimental): Patients with previously untreated, unresectable, locally advanced or metastatic GC/GEJ adenocarcinoma.
  Interventions: Drug: TST001; Drug: Nivolumab Injection [Opdivo]; Drug: mFOLFOX6
- Part B Cohort B (Experimental): Patients with GC/GEJ adenocarcinoma who have radiologically progressed following one or two prior systemic therapies.
  Interventions: Drug: TST001; Drug: Nivolumab Injection [Opdivo]
- Part B Cohort C (Experimental): Patients with previously untreated, unresectable, locally advanced or metastatic histologically confirmed pancreatic adenocarcinoma.
  Interventions: Drug: TST001; Drug: Gemcitabine; Drug: Albumin-Bound Paclitaxel

INTERVENTIONS:
Drug: TST001 — TST001 is a humanized IgG1 monoclonal antibody.
Drug: Nivolumab Injection [Opdivo] — Nivolumab is one of the PD-1 checkpoint inhibitors, and has proved clinical benefit for multiple late-stage malignancies
  Arms: Part B Cohort A; Part B Cohort B
Drug: mFOLFOX6 — mFOLFOX6 is a combination chemotherapy regimen including the drugs leucovorin calcium (folinic acid), fluorouracil, and oxaliplatin.
  Arms: Part B Cohort A
Drug: Gemcitabine — Chemotherapy medication
  Other Names: Gemzar
  Arms: Part B Cohort C
Drug: Albumin-Bound Paclitaxel — Chemotherapy medication
  Arms: Part B Cohort C

SUMMARY:
This is an open label Phase I/IIa, First in Human trial of TST001, a recombinant humanized anti-Claudin 18.2 (CLDN18.2) IgG1 monoclonal antibody as monotherapy or in combination with nivolumab or standard of care. It is being tested against advanced and/or metastatic solid tumors including gastric, gastroesophageal junction, pancreatic cancers.

DETAILED DESCRIPTION:
Part A of the trial will consist of two cohorts, one dosed every 2 weeks and one dosed every 3 weeks in a standard 3+3 design. Part A is the dose finding portion of the trial.

18 to 36 participants will be enrolled.

Part B consists of 3 cohorts:

Cohort A is for patients with previously untreated, unresectable, locally advanced or metastatic GC/GEJ adenocarcinoma. Patients will receive TST001 at 2mg/kg or 4mg/kg Q2W plus Nivolumab and mFOLFOX6. Alternative allocation of patients between the 2 doses will be performed. The first 6 patients at each dose level as the lead-in phase will not be selected on the basis of their tumor's CLDN18.2 expression. Approximately 12-42 patients will be enrolled in Cohort A.

Cohort B is for patients with GC/GEJ adenocarcinoma who have radiologically progressed following one or two prior systemic therapies. Patient will receive TST001 plus Nivolumab. No selection based on CLDN18.2 expression will be required for the safety run-in (3-6 patients). Patients with CLDN18.2 expression in tumor tissue tested by the central laboratory will be enrolled in the expansion phase. Safety run-in phase will follow 3+3 rule with two dose levels, TST001 3mg/kg and 6mg/kg Q3W combined with nivolumab. Approximately 30 patients will be enrolled in Cohort B including the patients in the safety run-in phase.

Cohort C is for patients with previously untreated, unresectable, locally advanced or metastatic histologically confirmed pancreatic adenocarcinoma; Patients will receive TST001 at 2mg/kg or 4mg/kg Q2W plus gemcitabine and albumin-bound paclitaxel. Alternative allocation of patients between the 2 doses will be performed. The first 6 patients at each dose level as the lead-in phase will not be selected on the basis of their tumor's CLDN18.2 expression. Approximately 12-42 patients will be enrolled in Cohort C.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 18 years.
* Patients with histologically or cytologically confirmed, locally advanced or metastatic solid tumors.

Part A only:

* Patients must be: a) progressed after standard therapies, b) intolerant of standard therapies, or c) with a tumor type without standard therapy.

Part B only:

* Cohort A: Patients with previously untreated, unresectable, locally advanced or metastatic GC/GEJ adenocarcinoma; prior adjuvant or neoadjuvant therapy are allowed only if disease progressed or recurred at least 6 months after completion of these treatments. Patients may have received one infusion of mFOLFOX6 plus nivolumab during the screening period.
* Cohort B: Patients with GC/GEJ adenocarcinoma who have radiologically progressed following one or two prior systemic therapies; adjuvant or neoadjuvant therapy could be regarded as one line of therapy only if disease progressed or recurred during these treatments or within 6 months or less after completion of these treatments.
* Cohort C: Patients with previously untreated, unresectable, locally advanced or metastatic histologically confirmed pancreatic adenocarcinoma; prior adjuvant or neoadjuvant therapy are allowed only if disease progressed or recurred at least 6 months after completion of these treatments. Patients may have received up to 2 infusions of Gemcitabine + albumin-bound paclitaxel (with one week between each infusion) during the screening period.
* Eastern Cooperative Oncology Group Performance Status (ECOG PS): 0-1 .
* Patients with adequate cardiac, liver, renal function, etc.

Exclusion Criteria

* Symptomatic central nervous system metastases.
* Prior treatment with any CLDN18.2 target agents
* Allergy or sensitivity to TST001 or known allergies to comparable drugs
* Documented history of multiple other allergies requiring interventions
* Severe cardiovascular disease, including CVA, TIA, myocardial infarction, or unstable angina, NYHA class III or IV heart failure or uncontrolled arrhythmia within 6 months of study entry, severe QTc prolongation, concomitant risks for QTc prolongation.
* Concurrent malignancy within 5 years prior to entry except adequately treated certain types of cancer
* Active and clinically significant infections, known uncontrolled infections with hepatitis B, hepatitis C, known human immunodeficiency virus with acquired immunodeficiency syndrome related illness
* Any condition that the investigator or primary physician believes may not be appropriate for participating in the study.

Other protocol-defined Inclusion/Exclusion Criteria could apply.

.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2020-05-28 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Participant Safety as characterized by frequency and severity of adverse events | up to 100 days following last dose
  Characterization of TST001 safety profile including frequency and severity of adverse events that are related to treatment.
Maximum Tolerated Dose (MTD or Recommended Phase 2 Dose (RP2D) | up to 100 days following last dose
  As measured by number of participants experiencing dose related toxicity (DLT) in each escalating cohort
Participant Safety and Tolerability of TST001 in combination with Nivolumab as characterized by frequency and severity of adverse events | Up to 100 days following last dose
  Characterization of TST001 + Nivolumab safety profile including frequency and severity of adverse events that are related to treatment.
Participant Safety and Tolerability of TST001 in combination with Nivolumab and mFOLFOX6 as characterized by frequency and severity of adverse events | Up to 100 days following last dose
  Characterization of TST001 + Nivolumab + mFOLFOX6 safety profile including frequency and severity of adverse events that are related to treatment.
Participant Safety and Tolerability of TST001 in combination with gemcitabine and albumin-bound paclitaxel as characterized by frequency and severity of adverse events | Up to 100 days following last dose
  Characterization of TST001 + Gemcitabine + albumin-bound paclitaxel safety profile including frequency and severity of adverse events that are related to treatment.

SECONDARY OUTCOMES:
Immunogenicity | up to 30 days following last dose
  by measurement of Incidence of anti-drug antibodies (ADA)
Objective response rate (ORR) | up to 24 months, until disease progression or start of another anti-cancer therapy
  as measured by RECIST 1.1
Duration of Response (DOR) | up to 24 months, until disease progression or start of another anti-cancer therapy
  duration of response (DOR)
Progression free survival (PFS) | up to 24 months, until disease progression or start of another anti-cancer therapy
  as measured by RECIST v1.1
PK parameters | Up to 30 days following last dose
  Maximum serum concentration (Cmax)
PK | Up to 30 days following last dose
  time to reach maximum serum concentration (Tmax)
PK | Up to 30 days following last dose
  Area Under the Curve

CONTACTS AND LOCATIONS:
Overall Officials: Charlie Qi, MD, Study Director — Suzhou Transcenta Therapeutics Co.
Locations (18):
- United States (18):
  - Banner MD Anderson, Gilbert, Arizona
  - University of Arizona, Tucson, Arizona
  - Yale University, New Haven, Connecticut
  - Florida Cancer Specialists, Sarasota, Florida
  - Emory University, Atlanta, Georgia
  - University of Kansas, School of Medicine, Kansas City, Kansas
  - Washington University, St Louis, Missouri
  - Memorial Sloan Kettering, New York, New York
  - Stony Brook Cancer Center, Stony Brook, New York
  - Wake Forest Baptist Comprehensive Cancer Center, Winston-Salem, North Carolina
  - Gabrail Cancer Research, Canton, Ohio
  - Pennsylvania Cancer Specialist Research Institute, Gettysburg, Pennsylvania
  - Allegheny Hospital, Pittsburgh, Pennsylvania
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Vanderbilt University, Nashville, Tennessee
  - NEXT Oncology, Austin, Texas
  - Swedish Cancer Institute, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
As described below. Patient personal data will be kept confidential as per HIPAA.
Supporting Information: Study Protocol, CSR
Time Frame: Clinical Study Report will become available approximately 60 to 90 days after last patient last visit. Each Investigator will receive one to keep. Protocol will be received prior to study start for each investigator.
Access Criteria: Be an active investigator in the TST001-1001 trial